CLINICAL TRIAL: NCT06491342
Title: PROBIOTIC SUPPLEMENT VERSUS PLACEBO FOR DECREASE STEATOSIS IN METABOLIC DYSFUNCTION-ASSOCIATED STEATOTIC LIVER DISEASE (MASLD): A MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED TRIAL
Brief Title: Probiotic Supplement Versus Placebo for the Treatment of Patients With Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Collaborators: Chiang Mai University (Other); Thailand Institute of scientific and technological research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMK GI 001
Record Dates: First submitted 2024-06-16; First posted 2024-07-09 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Fatty Liver, Nonalcoholic
Keywords: Probiotic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: probiotic vs placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin in bovine gelatin capsule look same as probiotic (250 mg/capsule ) 2 capsule twice daily after breakfast and dinner
  Interventions: Dietary Supplement: Placebo
- probiotic (Active Comparator): Lactobacillus Zeae and Lactobacillus reuteri probiotic mixed with Maltodextrin in ratio 15:85 in bovine gelatin capsule (250 mg/capsule ) 2 capsule twice daily after breakfast and dinner (1,000 mg =1x109 CFU/g)
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic-Lactobacillus Zeae and Lactobacillus reuteri
  Arms: probiotic
Dietary Supplement: Placebo — placebo
  Arms: Placebo

SUMMARY:
Probiotic supplement versus placebo for the treatment of patients with non-alcoholic fatty liver disease: a randomized, double-blind, placebo-controlled trial

DETAILED DESCRIPTION:
Probiotic supplement versus placebo for the treatment of patients with non-alcoholic fatty liver disease: a randomized, double-blind, placebo-controlled trial by access liver biochemistry, MRI-PDFF, fibroscan and metabolic profile

ELIGIBILITY:
Inclusion Criteria: Male and female adults ≥20,<80 years of age who suspected or confirmed diagnosis of NASH/NAFLD suggested by the historical data, they must meet one of the following criteria:

Fatty liver by imaging then fibroScan with CAP ≥ 248 dB m Liver biopsy compatible with NASH/NAFLD

Exclusion Criteria:

1. Supplement with probiotic/prebiotic within 2 weeks
2. Previous antibiotic/antifungus within 1 month
3. History of significant alcohol consumption for a period of more than three consecutive months within 1 year before screening. Significant alcohol consumption is defined as equal to or greater than approximately two alcoholic drinks per day for males and approximately 1.5 alcoholic drinks per day for females
4. Regular use of drugs historically associated with NAFLD, which include, but are not limited, to the following: amiodarone, methotrexate, systemic glucocorticoids at greater than 5 mg/d
5. Chronic liver diseases from other cause such as viral hepatitis, autoimmune hepatitis
6. Hepatic decompensation or impairment defined as presence of any of the following:

   * History of esophageal varices, ascites or hepatic encephalopathy.
   * Serum albumin <3.5 g dl-1, except as explained by nonhepatic causes.
   * INR > 1.4
7. Use of GLP-1 agonist therapy (for example, exenatide, liraglutide, lixisenatide, albiglutide, dulaglutide, semaglutide and albiglutide), vitamin E and pioglitazone
8. Active autoimmune disease, including actively treated lupus, rheumatoid arthritis, inflammatory bowel disease
9. Active malignancy on treatment
10. New York Heart Association Class III or IV heart failure or known left ventricular ejection fraction <30%
11. Known immunocompromised status, HIV or who have recurrent or chronic systemic bacterial, fungal, viral or protozoal infections
12. Respiratory compromised
13. Severe renal impairment (eGFR <30 ml/min/1.73 m2)
14. Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Liver steatosis by fibroscan | 12 weeks
  Shear wave velocity with controlled attenuation parameter (CAP) unit in decibels per meter (dB/m)
Liver steatosis by MRI | 12 weeks
  Hepatic steatosis with MRI-PDFF (the percent ratio of the density of mobile protons from triglycerides and the total density of protons from mobile triglycerides and mobile water). Outcome Measures was report as percent
Liver stiffness by fibroscan | 12 weeks
  Fibroscan- transient elastography in kilopascals (kPa)

SECONDARY OUTCOMES:
Liver inflammation | 12 weeks
  Evaluated alanine aminotransferase (ALT; U/L), aspartate aminotransferase (AST; U/L), gamma-glutamyl transferase (GGT; U/L), and alkaline phosphatase (ALP; U/L)
Metabolic profile | 12 weeks
  Fasting plasma glucose (FPG) in mg/dL
Metabolic profile | 12 weeks
  HbA1C in percent
Metabolic profile: HOMA IR | 12 weeks
  Fasting plasma glucose and serum insulin level will be combined to report in HOMA IR in mg/dl x mIU/L
Metabolic profile: serum lipid profiles | 12 weeks
  Total cholesterol in mg/dL, low-density lipoprotein (LDL) cholesterol in mg/dL, high-density lipoprotein (HDL) in mg/dl, cholesterol in mg/dL, and triglyceride in mg/dL
Inflammatory marker | 12 weeks
  hsCRP level in mg/L
Inflammatory marker | 12 weeks
  Interleukin 6 (IL-6) in pg/mL
Anthropomorphic evaluation: BMI | 12 weeks
  Weight and height will be combined to report BMI in kg/m^2
Anthropomorphic evaluation: composition analysis | 12 weeks
  Body fat in percentage
Anthropomorphic evaluation | 12 weeks
  Body muscle in kilogram

OTHER OUTCOMES:
Fecal SCFA | 12 weeks
  Fecal SCFA (acetate, propionate and butyrate) in microgram/ml metagenomic sequencing (Next-generation sequencing)

CONTACTS AND LOCATIONS:
Overall Officials: Natchaporn Noppacroh, Principal Investigator — phramongkutklao
Locations (2):
- Thailand (2):
  - Division of gastroenterology and hepatology, Ratchathewi, Bangkok
  - Chiangmai university, Chiang Mai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanyal AJ, Brunt EM, Kleiner DE, Kowdley KV, Chalasani N, Lavine JE, Ratziu V, McCullough A. Endpoints and clinical trial design for nonalcoholic steatohepatitis. Hepatology. 2011 Jul;54(1):344-53. doi: 10.1002/hep.24376. PMID 21520200
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Chang Y, Jung HS, Cho J, Zhang Y, Yun KE, Lazo M, Pastor-Barriuso R, Ahn J, Kim CW, Rampal S, Cainzos-Achirica M, Zhao D, Chung EC, Shin H, Guallar E, Ryu S. Metabolically Healthy Obesity and the Development of Nonalcoholic Fatty Liver Disease. Am J Gastroenterol. 2016 Aug;111(8):1133-40. doi: 10.1038/ajg.2016.178. Epub 2016 May 17. PMID 27185080
- [Background] Schnabl B, Brenner DA. Interactions between the intestinal microbiome and liver diseases. Gastroenterology. 2014 May;146(6):1513-24. doi: 10.1053/j.gastro.2014.01.020. Epub 2014 Jan 15. PMID 24440671
- [Background] Trinchieri G, Sher A. Cooperation of Toll-like receptor signals in innate immune defence. Nat Rev Immunol. 2007 Mar;7(3):179-90. doi: 10.1038/nri2038. PMID 17318230
- [Background] Imajo K, Fujita K, Yoneda M, Nozaki Y, Ogawa Y, Shinohara Y, Kato S, Mawatari H, Shibata W, Kitani H, Ikejima K, Kirikoshi H, Nakajima N, Saito S, Maeyama S, Watanabe S, Wada K, Nakajima A. Hyperresponsivity to low-dose endotoxin during progression to nonalcoholic steatohepatitis is regulated by leptin-mediated signaling. Cell Metab. 2012 Jul 3;16(1):44-54. doi: 10.1016/j.cmet.2012.05.012. PMID 22768838
- [Background] Wang S, Charbonnier LM, Noval Rivas M, Georgiev P, Li N, Gerber G, Bry L, Chatila TA. MyD88 Adaptor-Dependent Microbial Sensing by Regulatory T Cells Promotes Mucosal Tolerance and Enforces Commensalism. Immunity. 2015 Aug 18;43(2):289-303. doi: 10.1016/j.immuni.2015.06.014. Epub 2015 Jul 28. PMID 26231118
- [Background] Cani PD, Possemiers S, Van de Wiele T, Guiot Y, Everard A, Rottier O, Geurts L, Naslain D, Neyrinck A, Lambert DM, Muccioli GG, Delzenne NM. Changes in gut microbiota control inflammation in obese mice through a mechanism involving GLP-2-driven improvement of gut permeability. Gut. 2009 Aug;58(8):1091-103. doi: 10.1136/gut.2008.165886. Epub 2009 Feb 24. PMID 19240062
- [Background] Zhu L, Baker SS, Gill C, Liu W, Alkhouri R, Baker RD, Gill SR. Characterization of gut microbiomes in nonalcoholic steatohepatitis (NASH) patients: a connection between endogenous alcohol and NASH. Hepatology. 2013 Feb;57(2):601-9. doi: 10.1002/hep.26093. Epub 2013 Jan 8. PMID 23055155
- [Background] Bron PA, Kleerebezem M, Brummer RJ, Cani PD, Mercenier A, MacDonald TT, Garcia-Rodenas CL, Wells JM. Can probiotics modulate human disease by impacting intestinal barrier function? Br J Nutr. 2017 Jan;117(1):93-107. doi: 10.1017/S0007114516004037. PMID 28102115
- [Background] Alisi A, Bedogni G, Baviera G, Giorgio V, Porro E, Paris C, Giammaria P, Reali L, Anania F, Nobili V. Randomised clinical trial: The beneficial effects of VSL#3 in obese children with non-alcoholic steatohepatitis. Aliment Pharmacol Ther. 2014 Jun;39(11):1276-85. doi: 10.1111/apt.12758. Epub 2014 Apr 16. PMID 24738701
- [Background] Abhari K, Saadati S, Yari Z, Hosseini H, Hedayati M, Abhari S, Alavian SM, Hekmatdoost A. The effects of Bacillus coagulans supplementation in patients with non-alcoholic fatty liver disease: A randomized, placebo-controlled, clinical trial. Clin Nutr ESPEN. 2020 Oct;39:53-60. doi: 10.1016/j.clnesp.2020.06.020. Epub 2020 Jul 24. PMID 32859329
- [Background] Ferolla SM, Couto CA, Costa-Silva L, Armiliato GN, Pereira CA, Martins FS, Ferrari Mde L, Vilela EG, Torres HO, Cunha AS, Ferrari TC. Beneficial Effect of Synbiotic Supplementation on Hepatic Steatosis and Anthropometric Parameters, But Not on Gut Permeability in a Population with Nonalcoholic Steatohepatitis. Nutrients. 2016 Jun 28;8(7):397. doi: 10.3390/nu8070397. PMID 27367724
- [Background] Zhou D, Fan JG. Microbial metabolites in non-alcoholic fatty liver disease. World J Gastroenterol. 2019 May 7;25(17):2019-2028. doi: 10.3748/wjg.v25.i17.2019. PMID 31114130
- [Background] Rau M, Rehman A, Dittrich M, Groen AK, Hermanns HM, Seyfried F, Beyersdorf N, Dandekar T, Rosenstiel P, Geier A. Fecal SCFAs and SCFA-producing bacteria in gut microbiome of human NAFLD as a putative link to systemic T-cell activation and advanced disease. United European Gastroenterol J. 2018 Dec;6(10):1496-1507. doi: 10.1177/2050640618804444. Epub 2018 Sep 30. PMID 30574320
- [Background] Grundy SM, Cleeman JI, Daniels SR, Donato KA, Eckel RH, Franklin BA, Gordon DJ, Krauss RM, Savage PJ, Smith SC Jr, Spertus JA, Costa F; American Heart Association; National Heart, Lung, and Blood Institute. Diagnosis and management of the metabolic syndrome: an American Heart Association/National Heart, Lung, and Blood Institute Scientific Statement. Circulation. 2005 Oct 25;112(17):2735-52. doi: 10.1161/CIRCULATIONAHA.105.169404. Epub 2005 Sep 12. No abstract available. PMID 16157765
- [Background] Carr RM, Oranu A, Khungar V. Nonalcoholic Fatty Liver Disease: Pathophysiology and Management. Gastroenterol Clin North Am. 2016 Dec;45(4):639-652. doi: 10.1016/j.gtc.2016.07.003. Epub 2016 Oct 13. PMID 27837778
- [Background] Castera L, Friedrich-Rust M, Loomba R. Noninvasive Assessment of Liver Disease in Patients With Nonalcoholic Fatty Liver Disease. Gastroenterology. 2019 Apr;156(5):1264-1281.e4. doi: 10.1053/j.gastro.2018.12.036. Epub 2019 Jan 18. PMID 30660725
- [Background] Sasso M, Beaugrand M, de Ledinghen V, Douvin C, Marcellin P, Poupon R, Sandrin L, Miette V. Controlled attenuation parameter (CAP): a novel VCTE guided ultrasonic attenuation measurement for the evaluation of hepatic steatosis: preliminary study and validation in a cohort of patients with chronic liver disease from various causes. Ultrasound Med Biol. 2010 Nov;36(11):1825-35. doi: 10.1016/j.ultrasmedbio.2010.07.005. Epub 2010 Sep 27. PMID 20870345
- [Background] Dietrich CF, Bamber J, Berzigotti A, Bota S, Cantisani V, Castera L, Cosgrove D, Ferraioli G, Friedrich-Rust M, Gilja OH, Goertz RS, Karlas T, de Knegt R, de Ledinghen V, Piscaglia F, Procopet B, Saftoiu A, Sidhu PS, Sporea I, Thiele M. EFSUMB Guidelines and Recommendations on the Clinical Use of Liver Ultrasound Elastography, Update 2017 (Long Version). Ultraschall Med. 2017 Aug;38(4):e16-e47. doi: 10.1055/s-0043-103952. Epub 2017 Apr 13. PMID 28407655
- [Background] Shen QL, Chen YJ, Wang ZM, Zhang TC, Pang WB, Shu J, Peng CH. Assessment of liver fibrosis by Fibroscan as compared to liver biopsy in biliary atresia. World J Gastroenterol. 2015 Jun 14;21(22):6931-6. doi: 10.3748/wjg.v21.i22.6931. PMID 26078570
- [Background] Noureddin M, Lam J, Peterson MR, Middleton M, Hamilton G, Le TA, Bettencourt R, Changchien C, Brenner DA, Sirlin C, Loomba R. Utility of magnetic resonance imaging versus histology for quantifying changes in liver fat in nonalcoholic fatty liver disease trials. Hepatology. 2013 Dec;58(6):1930-40. doi: 10.1002/hep.26455. Epub 2013 Oct 17. PMID 23696515
- [Background] Middleton MS, Heba ER, Hooker CA, Bashir MR, Fowler KJ, Sandrasegaran K, Brunt EM, Kleiner DE, Doo E, Van Natta ML, Lavine JE, Neuschwander-Tetri BA, Sanyal A, Loomba R, Sirlin CB; NASH Clinical Research Network. Agreement Between Magnetic Resonance Imaging Proton Density Fat Fraction Measurements and Pathologist-Assigned Steatosis Grades of Liver Biopsies From Adults With Nonalcoholic Steatohepatitis. Gastroenterology. 2017 Sep;153(3):753-761. doi: 10.1053/j.gastro.2017.06.005. Epub 2017 Jun 15. PMID 28624576
- [Background] Ahn SB, Jun DW, Kang BK, Lim JH, Lim S, Chung MJ. Randomized, Double-blind, Placebo-controlled Study of a Multispecies Probiotic Mixture in Nonalcoholic Fatty Liver Disease. Sci Rep. 2019 Apr 5;9(1):5688. doi: 10.1038/s41598-019-42059-3. PMID 30952918
- [Background] Doron S, Snydman DR. Risk and safety of probiotics. Clin Infect Dis. 2015 May 15;60 Suppl 2(Suppl 2):S129-34. doi: 10.1093/cid/civ085. PMID 25922398
- [Background] Snydman DR. The safety of probiotics. Clin Infect Dis. 2008 Feb 1;46 Suppl 2:S104-11; discussion S144-51. doi: 10.1086/523331. PMID 18181712
- [Background] Salminen MK, Rautelin H, Tynkkynen S, Poussa T, Saxelin M, Valtonen V, Jarvinen A. Lactobacillus bacteremia, clinical significance, and patient outcome, with special focus on probiotic L. rhamnosus GG. Clin Infect Dis. 2004 Jan 1;38(1):62-9. doi: 10.1086/380455. Epub 2003 Dec 4. PMID 14679449
- [Background] Sullivan A, Nord CE. Probiotic lactobacilli and bacteraemia in Stockholm. Scand J Infect Dis. 2006;38(5):327-31. doi: 10.1080/00365540500449826. PMID 16709533
- [Background] Zielinska D, Sionek B, Kołozyn-Krajewska D. Safety of Probiotics. Diet, Microbiome and Health. 2018;:131-161
- [Background] Chambers ES, Viardot A, Psichas A, Morrison DJ, Murphy KG, Zac-Varghese SE, MacDougall K, Preston T, Tedford C, Finlayson GS, Blundell JE, Bell JD, Thomas EL, Mt-Isa S, Ashby D, Gibson GR, Kolida S, Dhillo WS, Bloom SR, Morley W, Clegg S, Frost G. Effects of targeted delivery of propionate to the human colon on appetite regulation, body weight maintenance and adiposity in overweight adults. Gut. 2015 Nov;64(11):1744-54. doi: 10.1136/gutjnl-2014-307913. Epub 2014 Dec 10. PMID 25500202
- [Background] Zhou D, Pan Q, Liu XL, Yang RX, Chen YW, Liu C, Fan JG. Clostridium butyricum B1 alleviates high-fat diet-induced steatohepatitis in mice via enterohepatic immunoregulation. J Gastroenterol Hepatol. 2017 Sep;32(9):1640-1648. doi: 10.1111/jgh.13742. PMID 28109017